CLINICAL TRIAL: NCT05482555
Title: Percutaneous Plug-based Femoral Arteriotomy Closure Device Use in Surgery for Acute Type A Aortic Disection
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Dalén, MD, PhD, Karolinska University Hospital
Other Study IDs: MANTA-ATAAD
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Aortic Dissection
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention/treatment Surgical cut-down and arterial puncture under direct vision: Surgical cut-down and arterial puncture under direct vision.
  Interventions: Procedure: Surgical cut-down and arterial puncture under direct vision
- Percutaneous arteriotomy closed with closure device: Percutaneous arteriotomy closed using a plug-based arteriotomy closure device (MANTA, Essential Medical Inc., Malvern, Pennsylvania).
  Interventions: Procedure: Percutaneous arteriotomy closed using a plug-based arteriotomy closure device

INTERVENTIONS:
Procedure: Percutaneous arteriotomy closed using a plug-based arteriotomy closure device — Percutaneous arteriotomy closed using a plug-based arteriotomy closure device (MANTA, Essential Medical Inc., Malvern, Pennsylvania).
  Groups: Percutaneous arteriotomy closed with closure device
Procedure: Surgical cut-down and arterial puncture under direct vision — Surgical cut-down and arterial puncture under direct vision.
  Groups: Intervention/treatment Surgical cut-down and arterial puncture under direct vision

SUMMARY:
A single-center prospective study. Patients undergoing surgery for acute type A aortic dissection with femoral arterial cannulation between 2017 and 2022 at the Karolinska University Hospital in Stockholm, Sweden are eligible. Femoral cannulation was performed either with surgical cut-down and arterial puncture under direct vision or percutaneously with planned percutaneous arteriotomy closed using a plug-based arteriotomy closure device (MANTA, Essential Medical Inc., Malvern, Pennsylvania). Data regarding preoperative clinical characteristics and operative details were obtained by medical records review.

ELIGIBILITY:
Inclusion Criteria:

* Operated for acute type A aortic dissection between 2017 and 2022 at the Karolinska University Hospital in Stockholm, Sweden.

Exclusion Criteria:

* Non-femoral arterial cannulation
* Concomitant femoro-femoral bypass
* Conversion to ECMO with arterial inflow in the previously cannulated femoral artery
* Death within 30 days from procedure
* Loss to follow-up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patientes operated for acute type A aortic dissection with femoral arterial cannulation between 2017 and 2022 at the Karolinska University Hospital in Stockholm, Sweden, with use of either surgical cut-down and arterial puncture under direct vision or percutaneously with planned percutaneous arteriotomy closed using a plug-based arteriotomy closure device.
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-06 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Femoral access site complication | During the first 8 weeks after surgery
  Seroma, wound infection, or nerve injury

SECONDARY OUTCOMES:
Femoral artery complication | During the first 3 years after surgery
  Pseudoaneurysm, local dissection, stenosis, intermittent claudication, or vascular closure device failure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiothoracic Surgery, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Individual participant data not planned to be shared.